CLINICAL TRIAL: NCT01506687
Title: Increasing Colorectal Cancer Screening Uptake With a Patient Navigator - Phase III Trial
Brief Title: Increasing Colorectal Cancer Screening Uptake With a Patient Navigator
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Care Ontario (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Paul Ritvo, Ph.D., Scientist, Research, Prevention and Cancer Control, Cancer Care Ontario
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 10-163
Record Dates: First submitted 2011-06-27; First posted 2012-01-10 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer screening; 50 years or older
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Navigator intervention (Experimental)
  Interventions: Behavioral: Health counselling by nurse navigator
- Usual Care Control (Active Comparator): Usual care
  Interventions: Behavioral: Usual primary care counselling

INTERVENTIONS:
Behavioral: Health counselling by nurse navigator — Information on colorectal cancer and screening, assistance in selection of screening option and obtaining kit or colonoscopy referral
  Other Names: Nurse navigator assistance
  Arms: Navigator intervention
Behavioral: Usual primary care counselling — Usual care health counselling on colorectal cancer and screening options
  Other Names: Usual primary care
  Arms: Usual Care Control

SUMMARY:
Patients who receive tailored navigation (consisting of a letter and patient navigation services) and get screened will be significantly greater than the control group who receives treatment as usual.

A majority of patients will opt for Fecal Occult Blood Testing (FOBT)as one of their preferred tests, after undergoing the "Patient Navigator" intervention and that proportion will be significantly greater than the group who opt for FOBT in the control group.

DETAILED DESCRIPTION:
Primary Outcome Measure:

Number of patients who receive a letter and patient navigation services and get screened compared to the control group.

Secondary Outcome Measures:

Proportion (%) of patients preferring FOBT vs.colonoscopy; Predictors of CRC screening and screening preference.

Subjects: Ambulatory patients (men-women aged 50 years and above) recruited from primary care practices at the Group Health Centre, Sault Ste Marie, Ontario. All patients will be screened for eligibility and those who are eligible and agree to participate in the study will be randomized to either of the two study arms: intervention group or control group.

ELIGIBILITY:
Inclusion Criteria:

* Average risk men and women aged 50 - 74
* Unscreened - Defined as no prior CRC screening
* Under-screened - Defined as no FOBT screening within the last two years
* No colonoscopy or barium enema screening within the last five years
* Willing to provide consent to participate in the study.

Exclusion Criteria:

* FOBT within the last two years
* colonoscopy within five years
* barium enema within five years
* flexible sigmoidoscopy within five years
* Bowel cancer.

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Completion of verified CRC screening event (FOBT;colonoscopy) event in experimental vs. control groups within 48 weeks | 48 weeks after baseline assessment
  Completion of verified CRC screening events in experimental vs. control patients

SECONDARY OUTCOMES:
Screening preferences; predictors of CRC screening and screening preference. | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul Ritvo, PHD, Principal Investigator — Cancer Care Ontario
Locations (1):
- Group Health Centre, Sault Ste. Marie, Ontario, Canada